CLINICAL TRIAL: NCT04592744
Title: Intraoperative Angiotensin 2 for the Prevention of Kidney Injury After Liver Transplant
Brief Title: Angiotensin 2 for AKI After OLT
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Colby Tanner, MD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-001402
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis, Liver; End Stage Liver DIsease; Acute Kidney Injury; Liver Transplant; Complications
MeSH Terms: conditions — Liver Cirrhosis; End Stage Liver Disease; Acute Kidney Injury | interventions — Angiotensin II; Norepinephrine; Vasopressins; Epinephrine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the intervention group receiving angiotensin 2 in addition to standard vasopressors or to the control group in which patients will receive standard vasopressors alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Patients assigned to the study group will receive Ang 2 infusion in addition to standard vasopressor regimen. Ang 2 is currently approved at UCLA as a second line vasopressor and will be used as such for the purposes of our study. Hemodynamic goals will be established at the beginning of the case by the anesthesiology and surgical teams. Ang 2 will be started as a second vasopressor once the norepinephrine dose has reached 0.05mcg/kg/min. Ang 2 will be initiated at a starting dose of 5ng/kg/min. That dose will be up titrated one time to 10ng/kg/min as vasopressor requirements escalate. Once a patient is on the 10ng/kg/min dose of ang 2, no additional up titration will be performed. Hemodynamic management will continue throughout the case with titration of other vasopressors as needed. Ang 2 will be continued throughout the intraoperative period but will be weaned off prior to leaving the operating room.
  Interventions: Drug: Angiotensin II; Drug: Norepinephrine
- Control (Active Comparator): Patients assigned to the control group will undergo intraoperative management with a standard vasopressor regimen composed of norepinephrine, vasopressin and epinephrine based on hemodynamic goals established by the surgical and anesthesia teams prior to surgery.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II infusion for Intraoperative management during liver transplantation
  Arms: Intervention
Drug: Norepinephrine — Vasopressor infusion for management of Intraoperative hypotension in liver transplantation.
  Other Names: Vasopressin; Epinephrine

SUMMARY:
Kidney injury is a common complication following liver transplantation and is associated with a higher complication rate and increased risk of death. While there are many factors that likely contribute to kidney injury in the perioperative period, a relative low serum level of angiotensin 2 (Ang 2) (a protein hormone that causes blood vessels to narrow) found in patients with liver cirrhosis (late stage of liver damage) may increase their risk of developing acute kidney injury (sudden episode of kidney failure or damage). We propose to investigate how early administration of Ang 2, a new vasopressor drug approved by the FDA in December 2017 for patients with low blood pressure, during the intra-operative period of liver transplant surgery affects the rate of kidney injury after transplantation. Patients who are deemed appropriate candidates for the study will be randomized 1:1 to the treatment and control groups. The intervention period of the study will occur in the operating room during transplant surgery and will be performed by their anesthesiologists. In the Treatment group, patients will receive Ang 2 infusions in addition to other standard vasopressors while patients in the control group will receive standard vasopressors alone. The infusion of Ang 2 in the treatment group will continue through the duration of the surgery and will be stopped prior to leaving the operating room. Both the treatment group and the control group will then be followed for 14 days to evaluate rates of kidney injury and to look for any complications. The follow up period will be extended to 28 days to look at in-hospital mortality rates in both groups. The daily follow up analysis will occur while the enrolled patients are inpatient following their transplantation surgery and will be done by looking at lab values and other data that is routinely gathered by their managing teams. This study will serve as a pilot study to evaluate feasibility of our protocol and to collect some preliminary data on the use of Ang 2 in this patient population. As such we plan to enroll approximately 30 patients who have accepted an offer to receive a donor liver. We hope to reach our goal enrollment within 5 months of starting the study.

DETAILED DESCRIPTION:
Acute kidney injury is a common perioperative complication following liver transplantation with an incidence of approximately 55%. Due to the complex physiologic derangements present in cirrhotic patients, multiple etiologies and processes may contribute, including chronic and acute hepatorenal syndrome, ATN, renal toxic medication administration, microvascular circulatory dysfunction from vasopressors, and hypoperfusion from the vasodilatory and hypovolemic forms of shock that are common during liver transplantation. While some of the risk factors for these causes of AKI can be mitigated, our current area of investigation revolves around the modulation of the renin-angiotensin system in the prevention of perioperative AKI. In cirrhosis, poor renal blood flow causes an increase in circulating levels plasma renin. However, recent studies suggest low levels of angiotensinogen and angiotensin 2, which are associated with AKI in cirrhotic patients5 and may contribute to the risk of perioperative AKI in liver transplant patients.

Angiotensin 2 was approved for clinical use as a vasopressor in 2017. The efficacy of angiotensin 2 at increasing systemic blood pressure in patients with vasodilatory shock was demonstrated by the ATHOS 3 trial. This study found that the addition of angiotensin 2 increased MAP by close to 10mmHg compared to placebo (12.5 vs 2.9 mmHg p< 0.001) and allowed for a decrease in other vasopressor utilization. Post-hoc analysis of the ATHOS-3 trial by Tumlin et al demonstrated that patients in vasodilatory shock with AKI had higher rates of recovery from AKI and fewer days requiring dialysis than those who did not receive angiotensin 2.

As vasodilatory shock is common among patients undergoing LT, this finding is relevant to our patient population. We hypothesize that angiotensin 2 will reduce AKI in patients undergoing LT, where vasodilatory shock is also very common.

Hypothesis: We propose that a relative deficiency of angiotensin 2 predisposes cirrhotic patients to develop acute kidney injury following liver transplantation. We hypothesize that initiating angiotensin 2 infusion as a short duration infusion during the intra-operative period of liver transplant surgery will decrease the incidence of postoperative acute kidney injury.

Aim1: Evaluate the efficacy of Angiotensin 2 to reduce incidence of acute kidney injury (AKI) following liver transplantation. Rates of recovery from AKI in patients with septic shock have been established in post-hoc analysis of the ATHOS-3 study. With high rates of AKI following transplant surgery as well as a patient population with predisposition for AKI in part due to a relative angiotensin 2 deficiency, we hope to demonstrate that the addition of angiotensin 2 to standard vasopressor regimens during transplant surgery decreases the incidence of postoperative AKI.

Aim 2: Evaluate the safety of angiotensin 2 in cirrhotic patients. While cirrhotic patients were included in the two largest studies of synthetic angiotensin 2 (ATHOS-1 and ATHOS-3), those with MELD > 40 were excluded, and no specific subgroup analysis was done. While several case reports of safe administration of angiotensin 2 in patients with cirrhosis have been published, we hope to further investigate its safety during liver transplant surgery. We hypothesize that angiotensin 2 can safely be administered in cirrhotic patients

ELIGIBILITY:
Inclusion Criteria:

A. End stage liver disease (ESLD) with acceptance of organ allocation offer. B. Stable renal function in the 48 hours prior to transplant (defined as < 30% change in serum creatinine) C. Adult patients > 18 years old

Exclusion Criteria:

A. Active use of renal replacement therapies B. Recent (within last 3 months) history of CVA or MI C. Patients with hypercoagulable state as evidenced by pre-existing venous thromboembolism or known thrombophilia (Antiphospholipid syndrome, Factor V- Leiden etc.) D. Combined liver transplant and intrathoracic surgery cases (not including chest tube placement) E. Multiple organ transplantation F. Congestive heart failure defined as left ventricular ejection fraction <45% G. Inability to obtain consent from the patient or surrogate H. Known allergy or sensitivity to any study medication I. Hepatocellular Carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute kidney Injury | Every day for 14 days following intervention
  Measured by change in serum creatinine from baseline based on KDIGO criteria.

SECONDARY OUTCOMES:
Need for Renal Replacement therapies | Every day for 14 days following intervention
In hospital mortalituy | 28 days
Urine output | 14 days
  Urine output measured in ml
Vasopressor doses | 14 days
  Vasopressor doses evaluated as norepinephrine equivalents
Adverse events | 14 days
  deep vein thrombosis, pulmonary embolus, intracardiac thrombus, stroke, myocardial infarction, peripheral ischemia, hepatic artery thrombosis, mesenteric ischemia, infusion site reaction, new infection, intraoperative tachycardia, intraoperative acidosis, lactatemia

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology & Perioperative Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Background] Tumlin JA, Murugan R, Deane AM, Ostermann M, Busse LW, Ham KR, Kashani K, Szerlip HM, Prowle JR, Bihorac A, Finkel KW, Zarbock A, Forni LG, Lynch SJ, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Bellomo R; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Outcomes in Patients with Vasodilatory Shock and Renal Replacement Therapy Treated with Intravenous Angiotensin II. Crit Care Med. 2018 Jun;46(6):949-957. doi: 10.1097/CCM.0000000000003092. PMID 29509568